CLINICAL TRIAL: NCT00625235
Title: The Use of a High Protein Diet in Achieving Long-Term Weight Loss and Improved Cardiovascular Risk Factors
Brief Title: A High Protein Diet and Weight Maintenance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Melbourne (Other)
Collaborators: Meat and Livestock Australia (Unknown)
Responsible Party: Meat and Livestock Australia
Allocation: Randomized | Model: Parallel | Purpose: Treatment
Other Study IDs: HREC 2003.046
Record Dates: First submitted 2008-02-19; First posted 2008-02-28 (Estimated); Last update posted 2008-02-28 (Estimated); Status verified 2003-06

CONDITIONS: Obesity
Keywords: Obesity; Weight loss; Weight maintenance; VLED
MeSH Terms: conditions — Obesity; Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Other): High Carbohydrate diet
  Interventions: Dietary Supplement: VLED followed by a high protein or high carbohydrate diet
- 2 (Other): High Protein diet
  Interventions: Dietary Supplement: VLED followed by a high protein or high carbohydrate diet

INTERVENTIONS:
Dietary Supplement: VLED followed by a high protein or high carbohydrate diet

SUMMARY:
An investigation into long term weight maintenance using a high protein or high carbohydrate diet, after a large and rapid weight loss.

ELIGIBILITY:
Inclusion Criteria:

* healthy men and women with a BMI >27kg/m2 with co-morbities or BMI >30kg/m2

Exclusion Criteria:

* people with Type II diabetes or other endocrine disorders, women who were pregnant or breastfeeding or planning to become pregnant

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180
Dates: Start 2003-07; Primary Completion 2006-01 (Actual); Study Completion 2006-01 (Actual)

PRIMARY OUTCOMES:
Body weight | 12 months

SECONDARY OUTCOMES:
Cardiovascular risk factors | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Medicine, Heidelberg Repatriation Hospital, Heidelberg, Victoria, Australia